CLINICAL TRIAL: NCT01968967
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled, Parallel-group Study To Assess The Efficacy, Long-term Safety And Tolerability Of Pf-04950615 In Subjects With Primary Hyperlipidemia Or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Brief Title: Randomized Clinical Trial of Bococizumab (PF-04950615; RN316) in Subjects With Hyperlipidemia or Mixed Dyslipidemia at Risk of Cardiovascular Events
Acronym: SPIRE-LDL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1481020; 2013-002643-28 (EudraCT Number); SPIRE-LDL (Other: Alias Study Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Hyperlipidemia
Keywords: mixed dyslipidemia; high risk of cardiovascular events; multiple cardiovascular disease risk factors
MeSH Terms: conditions — Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (PF-04950615; RN316) (Experimental)
  Interventions: Drug: Bococizumab (PF-04950615; RN316)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bococizumab (PF-04950615; RN316) — 150 mg every 2 weeks, subcutaneous injection, 12 months
  Arms: Bococizumab (PF-04950615; RN316)
Other: Placebo — subcutaneous injection every 2 weeks for 12 months
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized study in subjects with high cholesterol receiving highly effective statins to assess the efficacy, safety and tolerability of Bococizumab (PF-04950615;RN316) to lower LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a statin.
* Fasting LDL-C > 70 mg/dL and triglyceride <=400 mg/dL.
* High or very high risk of incurring a cardiovascular event.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* Cardiovascular or cerebrovascular event of procedures during the past 30 days.
* Congestive heart failure NYHA class IV.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2139 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (248):
- United States (154):
  - Ernest L. Hendrix, MD, PC, Athens, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - Alabama Internal Medicine, P.C., Birmingham, Alabama
  - Drug Shipment and Study Conducted at Address: University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, Llc, Huntsville, Alabama
  - Radiant Research Incorporated, Chandler, Arizona
  - Advanced Research Associates, Glendale, Arizona
  - Arizona Center For Internal Medicine, Mesa, Arizona
  - Holland Center for Family Health, Peoria, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Phoenix Clinical, Phoenix, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - Care Clinical Research Corporation, Banning, California
  - Med Center, Carmichael, California
  - Med Investigations, Fair Oaks, California
  - California Heart Specialists, Huntington Beach, California
  - Alia Clinical Research, Inc., Huntington Park, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Richard S. Cherlin, M.D., Los Gatos, California
  - California Medical Research Associates Inc., Northridge, California
  - Arch Health Partners Clinical Research Department, Poway, California
  - Clinical Trials Research, Sacramento, California
  - Northern California Research, Sacramento, California
  - Alta California Medical Group, Simi Valley, California
  - Orange County Research Center, Tustin, California
  - Empire Clinical Research, Upland, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Infosphere Clinical Research, INC, West Hills, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Clinical Research Advantage, Inc./Colorado Springs Health Partners, SW, Colorado Springs, Colorado
  - YNHH, Heart and Vascular, North Haven, Connecticut
  - ACRC-Cardiology, Atlantis, Florida
  - Morton Plant Mease Health Care, Inc. Cardiovascular Research, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - The Research Center, Inc., Hialeah, Florida
  - Homestead Medical Research Inc., Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, LLC at Baker-Gilmour Cardiovascular Institute, PA, Jacksonville, Florida
  - East Coast Institute for Research, LLC at Jacksonville Cardiovascular Center, Jacksonville, Florida
  - East Coast Institute for Research, LLC at Northeast Florida Cardiology Clinic, Jacksonville, Florida
  - East Coast Institute for Research, LLC at Northeast Florida Endocrine & Diabetes Associates, Jacksonville, Florida
  - St. Vincent's Cardiology, Jacksonville, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Clinical Research of Miami, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Medical Research Center, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Florida Institute For Clinical Research, LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - A&R Research Group, LLC, Pembroke Pines, Florida
  - DBC Research, Pembroke Pines, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - South Miami Clinical Research Center, LLC, South Miami, Florida
  - Dolphin Medical Research, Virginia Gardens, Florida
  - Metabolic Research Institute Incorporated, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Atlanta Center for Clinical Research / Internal Medicine, Roswell, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - American Health Network, LLC, Indianapolis, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - The University of Iowa - College of Public Health - Preventive Intervention Center, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Omega Clinical Research, Metairie, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Southern Maine Health Care, Biddeford, Maine
  - Columbia Medical Practice, Columbia, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - IHA Chelsea Family & Internal Medicine, Chelsea, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - Westside Family Medical Center, Pc, Kalamazoo, Michigan
  - Michigan Heart and Vascular Specialists, Petoskey, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - HealthEast St. Joseph's Hospital Pharmacy, Saint Paul, Minnesota
  - KCUMB Center for Community and Clinical Research, Kansas City, Missouri
  - Mercy Health Research, Washington, Missouri
  - Om Medical, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Rutgers Biomedical and Health Sciences- Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Premier Research, Trenton, New Jersey
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Drug Trials Brooklyn, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Crossroads Clinical Research, Inc., Mooresville, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Radiant Research, Inc, Akron, Ohio
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Sentral Clinical Research Services - Admin Only, Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - LION Research, Norman, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Detweiler Family Medicine and Associates, PC, Lansdale, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Warminster Medical Associates, P.C., Warminster, Pennsylvania
  - Coastal Cardiology, Charleston, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Cardiovascular Research of Knoxville, Knoxville, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - KRK Medical Research, Arlington, Texas
  - North Texas Healthcare System, Dallas VAMC, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - lnvestigational Drug Services (IDA), Houston, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Advanced Clinical Research Associates, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Bandera Family Health Care, LLC, San Antonio, Texas
  - Northwest Heart Center, Tomball, Texas
  - Radiant Research, Murray, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Amherst Family Practice, P.C., Winchester, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Zain Research LLC, Richland, Washington
- Canada (13):
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - Vizel Cardiac Research, Saul Vizel Professional Medicine Corporation, Cambridge, Ontario
  - The Office of Dr. Allen Greenspoon, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Stroke Prevention & Atherosclerosis Research Centre (SPARC), London, Ontario
  - Newmarket Cardiology Research Group, Newmarket, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - St. Michael's Hospital Health Centre, Toronto, Ontario
  - Rhodin Recherche Clinique, Drummondville, Quebec
  - LMC Research Inc. d.b.a. Manna Research Inc., Lévis, Quebec
  - Omnispec Clinical Research Inc., Mirabel, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - DIEX Research Sherbrooke Inc., Sherbrooke, Quebec
- Colombia (13):
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - Centro de Medicina del Ejercicio y Rehabilitacion Cardiaca S.A. CEMDE S.A., Medellín, Antioquia
  - Fundacion del Caribe para la Investigacion Biomedica-Fundacion Bios, Barranquilla, Atlántico
  - BIOMELAB Ltda., Barranquilla, Atlántico
  - IPS Centro Cientifico Asistencial Jose Luis Accini S.A.S., Barranquilla, Atlántico
  - Asociacion IPS Medicos InterniStas de Caldas, Manizales, Caldas Department
  - Dexa Diab Servicios Medicos Ltda. IPS, Bogota, Cundinamarca
  - Instituto de Investigacion Endocrinologia y Prevencion Metabolica ENDOCARE LTDA, Bogota, Cundinamarca
  - Centro de Diagnostico Cardiologico LTDA., Cartagena, Departamento de Bolívar
  - Fundacion Cardiomet - CEQUIN, Armenia, Quindío Department
  - Fundacion Cardiovascular De Colombia, Floridablanca, Santander Department
  - Fundacion Centro de Investigaciones Biomedicas RIESCARD, Espinal, Tolima Department
  - Centro de Investigaciones Clinicas S.A.S, Cali, Valle del Cauca Department
- France (5):
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU La Miletrie, Poitiers
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - Hopital Guy Chatiliez, Tourcoing
  - Hopital Guy Chatillez, Tourcoing
- Hungary (11):
  - Magyar Imre Korhaz, Belgyogyaszati Szakrendeles, Ajka
  - Bajai Szent Rokus Korhaz, Baja
  - Lausmed Kft., Baja
  - DRC Kft., Balatonfüred
  - SYNEXUS Magyarorszag Kft., Budapest
  - Synexus Magyarorzag Kft., Budapest
  - Pharma 4 Trial Kft., Gyöngyös
  - Borsod-Abauj-Zemplen Megyei Korhaz, es Egyetemi Oktatokorhaz, Miskolc
  - TaNaMed Kft., Mosonmagyaróvár
  - Pecsi Tudomanyegyetem, Pécs
  - Zala Megyei Korhaz, Zalaegerszeg
- Lithuania (4):
  - PI Kaunas Silainiai Outpatient Clinic, Kaunas
  - Private Clinic Elite Medicale, Kaunas
  - PI Klaipeda Seamen Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Mexico (10):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, S.C., Guadalajara, Jalisco
  - Clinicos Asociados BOCM, S.C., Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion S.C., Cuernavaca, Morelos
  - Administradora de Clinicas S.A. de C.V. Hospital Inovamed Cuernavaca, Cuernavaca, Morelos
  - Centro de Atención e Investigación Cardiovascular del Potosí S.C., San Luis Potosí City, San Luis Potosí
  - Hospital General de Naucalpan "Dr. Maximiliano Ruiz Castaneda" (Emergencies), Naucalpan, State of Mexico
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Centro de Investigacion Cardiometabolica de Aguascalientes SA de CV, Aguascalientes
  - Centro Hospitalario Mac, S.A. De C.V. (Emergencies), Aguascalientes
  - Hospital Angeles Centro Medico del Potosi (Emergencies), San Luis Potosí City
- Romania (5):
  - Spitalul Clinic Judetean de Urgenta Craiova, Cardiologie, Craiova, Dolj
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed, Medicina Interna, Brasov
  - Spitalul Universitar de Urgenta Militar Central, Dr. Carol Davila", Bucharest
  - Centrul Medical Unirea, Diabet Nutritie si Boli Metabolice, Cluj-Napoca
  - Elit Medical SRL, Ploieşti
- Russia (6):
  - Federal State Budgetary Institution "Research Institute of Complex problems of Cardio-vascular, Kemerovo
  - FSAEI of Higher Education "People's Friendship University of Russia",, Moscow
  - LLC "Institute of medical research", Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare Municipal hospital # 40 of the Kurortnyi, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare "Municipal Hospital #15", Saint Petersburg
  - Municipal Institution of Healthcare "City Clinical Hospital 12, Saratov
- Spain (9):
  - Centro Salud Petrer I, Petrel, Alicante
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario La Ribera, Alzira, Valencia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz; Unidad Metabolico-Vascular, Madrid
  - Hospital Clinico Universitario Miguel Servet; Medicina Interna, Zaragoza
- Taiwan (4):
  - Cardinal Tien Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (14):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Synexus Scotland Clinical Research Centre, Glasgow, Lanarkshire
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus Wales Clinical Research Centre, Cardiff, Llanishen
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - Northmed Clinical Research Ltd, Randalstown Health Centre, Antrim, Northern Ireland
  - Southern Health & Social Care Trust, Craigavon Area Hospital, Portadown, Northern Ireland
  - Synexus North East Clinical Research Centre-Hexham General Hospital, Hexham, Northumberland
  - Synexus North East Clinical Research Centre, Hexham, Northumberland
  - The Crouch Oak Family Practice, Addlestone, Surrey
  - Synexus Midlands Clinical Research Centre, Birmingham, WEST Midlands
  - The Bradford on Avon & Melksham Health Partnership, Bradford-on-Avon, Wiltshire
  - Ninewells Hospital & Medical School, Dundee

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] McCush F, Wang E, Yunis C, Schwartz P, Baltrukonis D. Anti-drug Antibody Magnitude and Clinical Relevance Using Signal to Noise (S/N): Bococizumab Case Study. AAPS J. 2023 Sep 2;25(5):85. doi: 10.1208/s12248-023-00846-x. PMID 37658997
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481020&StudyName=Randomized%20Clinical%20Trial%20of%20RN316%20%28PF-04950615%29%20in%20Subjects%20with%20Hyperlipidemia%20or%20Mixed%20Dyslipidemia%20at%20Risk%20of%20Cardiovascular%20Events

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at multiple sites from 28 October 2014 to 15 July 2016 for the Treatment Period and up to 10 July 2017 for the Extension Period.
Groups:
- Placebo (Treatment Period): Participants received placebo matched to Bococizumab (PF-04950615) subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
- Bococizumab 150 mg (Treatment Period): Participants received Bococizumab (PF-04950615) 150 milligram (mg) subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
- Placebo (Extension Period): Participants randomized to Placebo arm in treatment period and consented for extension period after Week 58 follow-up visit, were followed for SAEs and concomitant medications up to Week 110.
- Bococizumab ADA Positive (Extension Period): Participants randomized to Bococizumab in treatment period were classified as either ADA positive or ADA negative based on their ADA assessment at Week 58 follow-up visit. In extension period, participants who were ADA positive and consented for extension period were assessed for ADA and LDL-C direct measurement until ADA titers were no longer detectable or had returned to baseline titer (less than or equal to 1.58 (log2) units above a positive baseline titer) or until Week 110 along with SAEs and concomitant medication, from Week 58 follow up visit to Week 110.
- Bococizumab ADA Negative (Extension Period): Participants randomized to Bococizumab in treatment period were classified as either ADA positive or ADA negative based on their Week 58 follow-up ADA assessment. Participants who were ADA negative and consented for extension period were followed for SAEs and concomitant medication, from Week 58 follow up visit to Week 110.
Period: Treatment Period
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period) | Placebo (Extension Period) | Bococizumab ADA Positive (Extension Period) | Bococizumab ADA Negative (Extension Period)
Started | 1071 | 1068 | 0 | 0 | 0
Treated | 1065 | 1063 | 0 | 0 | 0
Completed | 925 | 934 | 0 | 0 | 0
Not Completed | 146 | 134 | 0 | 0 | 0
Not completed — Other | 22 | 22 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 71 | 61 | 0 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 26 | 31 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 8 | 0 | 0 | 0
Not completed — Death | 9 | 2 | 0 | 0 | 0
Not completed — Randomized Not Treated | 6 | 5 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period) | Placebo (Extension Period) | Bococizumab ADA Positive (Extension Period) | Bococizumab ADA Negative (Extension Period)
Started | 0 | 0 | 47 | 19 | 39
Completed | 0 | 0 | 45 | 19 | 34
Not Completed | 0 | 0 | 2 | 0 | 5
Not completed — Withdrew Consent | 0 | 0 | 2 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Bococizumab 150 mg (Treatment Period): Participants received Bococizumab (PF--04950615) 150 mg subcutaneous injection once every 2 weeks up to Week 52 and were followed up to Week 58.
- Total: Total of all reporting groups
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period) | Total
Number analyzed (Participants) | 1071 | 1068 | 2139
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.8) | 61.8 (9.3) | 62 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 434 | 434 | 868
  Male | 637 | 634 | 1271

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, "Number of participants analyzed (N)" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Bococizumab 150 mg (Treatment Period): Participants received Bococizumab (PF--04950615) 150 mg subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 994 | 980
percent change | 1.0 (22.55) | -54.9 (26.84)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Least square (LS) mean difference and associated 95 percent (%) confidence interval (CI), and p-value were derived from mixed effect model repeat measurement (MMRM) model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -56.2, 95% CI 2-sided [-58.3 to -54.0], Standard Error of Mean 1.10

2. Secondary Outcome: Percent Change From Baseline in Fasting Total Cholesterol (TC) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 997 | 981
  Week 12 | -0.1 (16.18) | -34.9 (18.34)
  Week 24: number analyzed (Participants) | 988 | 988
  Week 24 | 1.0 (18.68) | -30.5 (21.56)
  Week 52: number analyzed (Participants) | 920 | 932
  Week 52 | -0.3 (18.75) | -25.3 (23.43)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 12: LS mean difference and associated 95% CI and p-value were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -35.0, 95% CI 2-sided [-36.5 to -33.5], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 24: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -31.6, 95% CI 2-sided [-33.3 to -29.8], Standard Error of Mean 0.89
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 52: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -24.7, 95% CI 2-sided [-26.6 to -22.8], Standard Error of Mean 0.96

3. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B (ApoB) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 994 | 978
  Week 12 | 0.4 (18.83) | -50.4 (27.42)
  Week 24: number analyzed (Participants) | 987 | 988
  Week 24 | 1.5 (21.43) | -44.9 (31.17)
  Week 52: number analyzed (Participants) | 915 | 929
  Week 52 | -0.4 (21.78) | -37.4 (32.92)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -50.8, 95% CI 2-sided [-52.9 to -48.8], Standard Error of Mean 1.04
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -46.1, 95% CI 2-sided [-48.5 to -43.8], Standard Error of Mean 1.19
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -36.1, 95% CI 2-sided [-38.6 to -33.6], Standard Error of Mean 1.28

4. Secondary Outcome: Percent Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 996 | 980
  Week 12 | 0.2 (21.22) | -49.7 (25.51)
  Week 24: number analyzed (Participants) | 987 | 987
  Week 24 | 1.6 (24.65) | -43.8 (30.02)
  Week 52: number analyzed (Participants) | 919 | 932
  Week 52 | -0.3 (24.62) | -36.8 (32.73)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -50.1, 95% CI 2-sided [-52.1 to -48.0], Standard Error of Mean 1.04
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -45.5, 95% CI 2-sided [-47.9 to -43.1], Standard Error of Mean 1.22
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -35.9, 95% CI 2-sided [-38.5 to -33.3], Standard Error of Mean 1.33

5. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides (TG) Cut-off of Less Than (<) 200 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: A subset of FAS included all participants who were randomized and had TG <200 mg/dL at pre-randomization. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 791 | 788
percent change
  Week 12: number analyzed (Participants) | 734 | 725
  Week 12 | 1.9 (23.07) | -55.6 (26.81)
  Week 24: number analyzed (Participants) | 730 | 729
  Week 24 | 3.9 (27.17) | -49.2 (32.58)
  Week 52: number analyzed (Participants) | 683 | 688
  Week 52 | 3.2 (26.65) | -40.6 (36.45)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 12: LS mean difference and associated 95% CI and p-value were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -57.7, 95% CI 2-sided [-60.2 to -55.2], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 24: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -53.1, 95% CI 2-sided [-56.1 to -50.0], Standard Error of Mean 1.55
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 52: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -42.8, 95% CI 2-sided [-46.2 to -39.5], Standard Error of Mean 1.70

6. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Greater Than or Equal to (>=) 200 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: A subset of FAS included all participants who were randomized and had TG >=200 mg/dL at pre-randomization. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 280 | 280
percent change
  Week 12: number analyzed (Participants) | 260 | 255
  Week 12 | -1.5 (20.82) | -53.0 (26.90)
  Week 24: number analyzed (Participants) | 257 | 260
  Week 24 | 1.1 (28.21) | -42.8 (31.87)
  Week 52: number analyzed (Participants) | 237 | 241
  Week 52 | -1.2 (27.78) | -36.3 (34.88)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -51.8, 95% CI 2-sided [-55.9 to -47.7], Standard Error of Mean 2.09
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 24: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -44.0, 95% CI 2-sided [-49.1 to -38.8], Standard Error of Mean 2.61
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 52: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -34.6, 95% CI 2-sided [-40.2 to -29.0], Standard Error of Mean 2.83

7. Secondary Outcome: Percent Change From Baseline in Fasting Lipoprotein (a) (Lp[a]) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 994 | 975
  Week 12 | 2.4 (85.08) | -26.3 (42.63)
  Week 24: number analyzed (Participants) | 984 | 983
  Week 24 | 8.7 (146.00) | -22.7 (51.48)
  Week 52: number analyzed (Participants) | 918 | 927
  Week 52 | 4.3 (139.49) | -20.9 (110.14)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -28.5, 95% CI 2-sided [-34.4 to -22.5], Standard Error of Mean 3.04
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -31.1, 95% CI 2-sided [-40.6 to -21.5], Standard Error of Mean 4.86
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -25.3, 95% CI 2-sided [-36.8 to -13.7], Standard Error of Mean 5.89

8. Secondary Outcome: Percent Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 996 | 981
  Week 12 | 0.4 (13.92) | 6.2 (14.99)
  Week 24: number analyzed (Participants) | 987 | 987
  Week 24 | 0.5 (15.25) | 6.1 (15.32)
  Week 52: number analyzed (Participants) | 919 | 932
  Week 52 | 1.2 (16.09) | 6.5 (17.87)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = 5.8, 95% CI 2-sided [4.5 to 7.0], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 5.5, 95% CI 2-sided [4.2 to 6.8], Standard Error of Mean 0.67
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = 5.2, 95% CI 2-sided [3.7 to 6.7], Standard Error of Mean 0.76

9. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 24, 52: Treatment Period
Time Frame: Baseline, Week 24, 52
Population: FAS included all participants who were randomized. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 24: number analyzed (Participants) | 987 | 989
  Week 24 | 3.2 (27.45) | -47.5 (32.50)
  Week 52: number analyzed (Participants) | 920 | 929
  Week 52 | 2.1 (27.00) | -39.5 (36.08)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -50.7, 95% CI 2-sided [-53.3 to -48.0], Standard Error of Mean 1.34
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -40.7, 95% CI 2-sided [-43.5 to -37.8], Standard Error of Mean 1.46

10. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 997 | 981
  Week 12 | 3.5 (38.25) | -12.9 (39.99)
  Week 24: number analyzed (Participants) | 988 | 988
  Week 24 | 5.1 (51.06) | -11.5 (41.33)
  Week 52: number analyzed (Participants) | 920 | 932
  Week 52 | 0.3 (43.63) | -12.5 (40.82)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 12: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -16.6, 95% CI 2-sided [-20.0 to -13.2], Standard Error of Mean 1.73
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -16.7, 95% CI 2-sided [-20.7 to -12.6], Standard Error of Mean 2.05
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -12.8, 95% CI 2-sided [-16.5 to -9.0], Standard Error of Mean 1.91

11. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 995 | 980
  Week 12 | -0.6 (11.22) | 2.8 (11.73)
  Week 24: number analyzed (Participants) | 987 | 988
  Week 24 | -0.9 (12.10) | 2.7 (11.93)
  Week 52: number analyzed (Participants) | 916 | 929
  Week 52 | -1.2 (12.34) | 2.6 (13.75)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 3.4, 95% CI 2-sided [2.4 to 4.3], Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 3.5, 95% CI 2-sided [2.5 to 4.5], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = 3.8, 95% CI 2-sided [2.7 to 4.9], Standard Error of Mean 0.57

12. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-II (ApoA-II) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 993 | 972
  Week 12 | -1.2 (13.05) | -1.0 (13.75)
  Week 24: number analyzed (Participants) | 986 | 986
  Week 24 | -0.9 (13.56) | 0.1 (14.28)
  Week 52: number analyzed (Participants) | 916 | 928
  Week 52 | -2.5 (13.50) | -1.0 (13.72)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.3, 95% CI 2-sided [-0.9 to 1.4], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 1.1, 95% CI 2-sided [-0.1 to 2.3], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = 1.5, 95% CI 2-sided [0.3 to 2.7], Standard Error of Mean 0.61

13. Secondary Outcome: Percent Change From Baseline in Fasting Very Low Density Lipoprotein Cholesterol (VLDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percent change
  Week 12: number analyzed (Participants) | 997 | 981
  Week 12 | 3.5 (38.25) | -12.9 (39.99)
  Week 24: number analyzed (Participants) | 988 | 988
  Week 24 | 5.1 (51.06) | -11.5 (41.33)
  Week 52: number analyzed (Participants) | 920 | 932
  Week 52 | 0.3 (43.63) | -12.5 (40.82)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -16.6, 95% CI 2-sided [-20.0 to -13.2], Standard Error of Mean 1.73
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -16.7, 95% CI 2-sided [-20.7 to -12.6], Standard Error of Mean 2.05
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -12.8, 95% CI 2-sided [-16.5 to -9.0], Standard Error of Mean 1.91

14. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Less Than (<) 200 Milligram Per Deciliter (mg/dL) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 791 | 788
mg/dL
  Baseline: number analyzed (Participants) | 791 | 787
  Baseline | 109.1 (33.24) | 107.1 (30.43)
  Change at Week 12: number analyzed (Participants) | 734 | 725
  Change at Week 12 | 0.3 (25.70) | -59.3 (32.30)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -60.4, 95% CI 2-sided [-63.1 to -57.6], Standard Error of Mean 1.40

15. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Greater Than or Equal to (>=) 200 Milligram Per Deciliter (mg/dL) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 280 | 280
mg/dL
  Baseline | 125.9 (40.08) | 121.5 (37.84)
  Change at Week 12: number analyzed (Participants) | 260 | 255
  Change at Week 12 | -3.4 (29.08) | -64.8 (38.94)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -62.8, 95% CI 2-sided [-68.3 to -57.3], Standard Error of Mean 2.80

16. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1071 | 1067
  Baseline | 113.5 (35.90) | 110.9 (33.13)
  Change at Week 12: number analyzed (Participants) | 994 | 980
  Change at Week 12 | -0.7 (26.66) | -60.7 (34.22)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -61.0, 95% CI 2-sided [-63.5 to -58.5], Standard Error of Mean 1.27

17. Secondary Outcome: Absolute Change From Baseline in Fasting Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1071 | 1067
  Baseline | 186.3 (40.77) | 183.1 (38.31)
  Change at Week 12: number analyzed (Participants) | 997 | 981
  Change at Week 12 | -1.8 (31.62) | -64.5 (38.01)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -63.7, 95% CI 2-sided [-66.6 to -60.9], Standard Error of Mean 1.46

18. Secondary Outcome: Absolute Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1071 | 1066
  Baseline | 138.0 (39.67) | 135.3 (36.85)
  Change at Week 12: number analyzed (Participants) | 996 | 980
  Change at Week 12 | -1.6 (30.93) | -67.0 (38.89)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -66.4, 95% CI 2-sided [-69.3 to -63.6], Standard Error of Mean 1.46

19. Secondary Outcome: Absolute Change From Baseline in Fasting Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1070 | 1067
  Baseline | 94.0 (24.26) | 92.3 (22.74)
  Change at Week 12: number analyzed (Participants) | 994 | 978
  Change at Week 12 | -0.7 (18.35) | -46.0 (26.58)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -45.8, 95% CI 2-sided [-47.7 to -43.9], Standard Error of Mean 0.97

20. Secondary Outcome: Absolute Change From Baseline in Fasting Lipoprotein (a) (Lp[a]) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1069 | 1063
  Baseline | 45.3 (49.77) | 46.4 (55.57)
  Change at Week 12: number analyzed (Participants) | 994 | 975
  Change at Week 12 | -0.0 (12.07) | -10.6 (18.36)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -10.6, 95% CI 2-sided [-11.8 to -9.3], Standard Error of Mean 0.63

21. Secondary Outcome: Absolute Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
mg/dL
  Baseline: number analyzed (Participants) | 1071 | 1066
  Baseline | 48.3 (12.42) | 47.8 (12.72)
  Change at Week 12: number analyzed (Participants) | 996 | 981
  Change at Week 12 | -0.1 (6.84) | 2.5 (7.07)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 2.7, 95% CI 2-sided [2.1 to 3.3], Standard Error of Mean 0.31

22. Secondary Outcome: Absolute Change From Baseline in Ratio of Fasting Total Cholesterol (TC) to High Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
Ratio
  Baseline: number analyzed (Participants) | 1071 | 1066
  Baseline | 4.1 (1.22) | 4.0 (1.19)
  Change at Week 12: number analyzed (Participants) | 996 | 980
  Change at Week 12 | -0.0 (0.86) | -1.5 (1.09)
  Change at Week 24: number analyzed (Participants) | 987 | 987
  Change at Week 24 | 0.0 (0.96) | -1.4 (1.15)
  Change at Week 52: number analyzed (Participants) | 919 | 932
  Change at Week 52 | -0.0 (0.97) | -1.1 (1.21)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -1.6, 95% CI 2-sided [-1.6 to -1.5], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -1.4, 95% CI 2-sided [-1.5 to -1.3], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -1.1, 95% CI 2-sided [-1.2 to -1.0], Standard Error of Mean 0.05

23. Secondary Outcome: Change From Baseline in Ratio of Fasting Apolipoprotein B (ApoB) to Apolipoprotein A-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
Ratio
  Baseline: number analyzed (Participants) | 1070 | 1067
  Baseline | 0.7 (0.21) | 0.7 (0.20)
  Change at Week 12: number analyzed (Participants) | 994 | 978
  Change at Week 12 | 0.0 (0.14) | -0.3 (0.21)
  Change at Week 24: number analyzed (Participants) | 987 | 988
  Change at Week 24 | 0.0 (0.15) | -0.3 (0.23)
  Change at Week 52: number analyzed (Participants) | 915 | 929
  Change at Week 52 | 0.0 (0.16) | -0.2 (0.23)
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 12: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -0.3, 95% CI 2-sided [-0.3 to -0.3], Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 24: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -0.3, 95% CI 2-sided [-0.3 to -0.3], Standard Error of Mean 0.01
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 52: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS Mean Difference = -0.2, 95% CI 2-sided [-0.3 to -0.2], Standard Error of Mean 0.01

24. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 100 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time points for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percentage of participants
  Week 12: number analyzed (Participants) | 994 | 980
  Week 12 | 45.3 | 90.9
  Week 2: number analyzed (Participants) | 987 | 990
  Week 2 | 43.2 | 85.8
  Week 52: number analyzed (Participants) | 920 | 930
  Week 52 | 45.0 | 79.8
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 12: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 27.0, 95% CI 2-sided [19.21 to 38.02]
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 24: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 12.9, 95% CI 2-sided [9.84 to 16.86]
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); Week 52: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 6.3, 95% CI 2-sided [4.99 to 8.06]

25. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 70 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1071 | 1068
percentage of participants
  Week 12: number analyzed (Participants) | 994 | 980
  Week 12 | 5.9 | 78.6
  Week 24: number analyzed (Participants) | 987 | 990
  Week 24 | 7.8 | 69.8
  Week 52: number analyzed (Participants) | 920 | 930
  Week 52 | 6.8 | 61.4
Statistical Analysis 1: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 86.5, 95% CI 2-sided [61.74 to 121.25]
Statistical Analysis 2: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 24, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 35.9, 95% CI 2-sided [26.83 to 47.96]
Statistical Analysis 3: Comparison: Placebo (Treatment Period) vs Bococizumab 150 mg (Treatment Period); [analysis description as in outcome 24, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 25.5, 95% CI 2-sided [18.90 to 34.47]

26. Secondary Outcome: Plasma Concentration of PF-04950615 at Week 12, 24 and 52
Description: Plasma concentration of PF-04950615 at Week 12, 24 and 52 was reported.
Time Frame: Week 12, 24, 52
Population: Analysis set included participants who received at least 1 dose of PF-04950615. Here, "n" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1063
Microgram per milliliter
  Week 12: number analyzed (Participants) | 996
  Week 12 | 4.91 (4.987)
  Week 24: number analyzed (Participants) | 975
  Week 24 | 4.74 (5.772)
  Week 52: number analyzed (Participants) | 915
  Week 52 | 3.60 (4.685)

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) Related to Type 1 or 3 Hypersensitivity Reactions and Injection Site Reactions
Description: Type 1 hypersensitivity or allergic reactions were possible in response to any injected protein and included shortness of breath, urticaria, anaphylaxis and angioedema. Type 3 hypersensitivity reactions were similar to Type 1 hypersensitivity reactions but were likely to be delayed from the time of injection and included symptoms such as rash, urticaria, polyarthritis, myalgia's, polysynovitis, fever and if severe then included glomerulonephritis. Injection site reactions included injection site bruising, discolouration, erythema, haematoma, haemorrhage, nodule, induration, inflammation, mass, pain, paraesthesia, pruritus, swelling, vesicles, warmth, scab and rash. Participants with type 1 or type 3 hypersensitivity reactions and participants with injection site reactions were reported in this outcome measure.
Time Frame: Baseline up to Week 58
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 1065 | 1063
Participants
  Type 1 or 3 hypersensitivity reactions | 2 | 2
  Injection site reactions | 56 | 144

28. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb): Treatment Period
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported. ADA titer >=6.23 (log2) unit was considered to be ADA positive and nAb titer >=1.58 (log2) unit was considered to be nAb positive.
Time Frame: Baseline up to Week 58
Population: Safety analysis population included all participants who received at least 1 dose of study treatment. Here, "N" signifies those participants who were evaluable for this outcome measure for each reporting arm respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period)
Number analyzed (Participants) | 231 | 1046
Percentage of participants
  Baseline up to Week 58: ADA | 0.9 | 46.7
  Baseline up to Week 58: nAb | 0.4 | 30.3

29. Secondary Outcome: Number of Participants Who Changed Concomitant Medication During Extension Period
Description: In this outcome measure, total number of participants who changed their lipid-lowering medications or added a monoclonal antibody medication during the extension period were reported.
Time Frame: Week 58 follow-up visit to Week 110
Population: All participants who consented for extension period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Extension Period) | Bococizumab ADA Positive (Extension Period) | Bococizumab ADA Negative (Extension Period)
Number analyzed (Participants) | 47 | 19 | 39
Participants | 2 | 1 | 2

30. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 58 Follow-up Visit, 71, 84, 97 and 110: Extension Period
Time Frame: Baseline, Week 58 follow-up visit, 71, 84, 97, 110
Population: All participants who consented for extension period. This outcome measure was planned not to be analyzed for reporting arms: Placebo (Extension Period) and Bococizumab ADA negative (Extension Period). Here, "n" signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Bococizumab ADA Positive (Extension Period)
Number analyzed (Participants) | 19
percent change
  Week 58 follow-up visit | -6.4 (24.67)
  Week 71: number analyzed (Participants) | 16
  Week 71 | -10.4 (41.51)
  Week 84: number analyzed (Participants) | 11
  Week 84 | -15.8 (25.65)
  Week 97: number analyzed (Participants) | 9
  Week 97 | -20.8 (31.08)
  Week 110: number analyzed (Participants) | 9
  Week 110 | -5.0 (28.65)

31. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb): Extension Period
Description: as for outcome 28
Time Frame: Week 58 follow-up visit, Week 71, Week 84, Week 97, Week 110
Population: All participants who consented for extension period. This outcome measure was planned not to be analyzed for reporting arms Placebo (Extension period) and Bococizumab ADA negative (Extension period). Here, "n" signifies number of participants who were evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Bococizumab ADA Positive (Extension Period)
Number analyzed (Participants) | 19
Percentage of participants
  Week 58 follow-up visit: ADA | 100.0
  Week 58 follow-up visit: nAB | 36.8
  Week 71: ADA: number analyzed (Participants) | 16
  Week 71: ADA | 62.5
  Week 71: nAB: number analyzed (Participants) | 16
  Week 71: nAB | 31.3
  Week 84: ADA: number analyzed (Participants) | 11
  Week 84: ADA | 81.8
  Week 84: nAB: number analyzed (Participants) | 11
  Week 84: nAB | 45.5
  Week 97: ADA: number analyzed (Participants) | 4
  Week 97: ADA | 50.0
  Week 97: nAB: number analyzed (Participants) | 4
  Week 97: nAB | 0.0
  Week 110: ADA: number analyzed (Participants) | 7
  Week 110: ADA | 85.7
  Week 110: nAB: number analyzed (Participants) | 7
  Week 110: nAB | 57.1

ADVERSE EVENTS:
Time Frame: For SAEs: Baseline up to Week 110 and for other AEs: Baseline up to Week 58
Description: Event may be serious in 1 and nonserious in other participant or 1 participant may have experienced both serious and nonserious AE. Participants evaluable:treatment period: participants who received at least 1 dose of study drug;extension period: participants who consented for extension period. Nonserious AEs were not collected for extension period.
Arm/Group | Placebo (Treatment Period) | Bococizumab 150 mg (Treatment Period) | Placebo (Extension Period) | Bococizumab ADA Positive (Extension Period) | Bococizumab ADA Negative (Extension Period)
All-Cause Mortality (participants affected / at risk) | 9/1065 | 2/1063 | 0/47 | 0/19 | 0/39
Serious Adverse Events (participants affected / at risk) | 150/1065 | 116/1063 | 1/47 | 1/19 | 1/39
Other Adverse Events (participants affected / at risk) | 138/1065 | 177/1063 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (Treatment Period) (N=1065) | Bococizumab 150 mg (Treatment Period) (N=1063) | Placebo (Extension Period) (N=47) | Bococizumab ADA Positive (Extension Period) (N=19) | Bococizumab ADA Negative (Extension Period) (N=39)
Left leg - severe pain, redness, and induration (General disorders) | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 7 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 4 | 8 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 6 | 2 | 0 | 0 | 0
Aortic valve calcification (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 4 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 4 | 3 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 4 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 3 | 0 | 0 | 0
Subvalvular aortic stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 2 | 0 | 0 | 0
Bartter's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 7 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 4 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1/635 | 0/630 | 0/31 | 0/8 | 0/26 — This event was gender specific.
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diabetic gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 3 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 1/635 | 0/630 | 0/31 | 0/8 | 0/26 — This event was gender specific.
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 0 | 0 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/430 | 1/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/430 | 1/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/430 | 0/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/635 | 0/630 | 0/31 | 0/8 | 0/26 — This event was gender specific.
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/430 | 0/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/430 | 1/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 3 | 0 | 0 | 0
Syncope (Nervous system disorders) | 8 | 2 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0/635 | 1/630 | 0/31 | 0/8 | 0/26 — This event was gender specific.
Scrotal ulcer (Reproductive system and breast disorders) | 1/635 | 0/630 | 0/31 | 0/8 | 0/26 — This event was gender specific.
Vaginal prolapse (Reproductive system and breast disorders) | 1/430 | 0/433 | 0/16 | 0/11 | 0/13 — This event was gender specific.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 4 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Condition aggravated (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Treatment Period) (N=1065) | Bococizumab 150 mg (Treatment Period) (N=1063) | Placebo (Extension Period) (N=0) | Bococizumab ADA Positive (Extension Period) (N=0) | Bococizumab ADA Negative (Extension Period) (N=0)
Injection site reaction (General disorders) | 23 | 97 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 60 | 50 | 0 | 0 | 0
Hypertension (Vascular disorders) | 61 | 47 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.